CLINICAL TRIAL: NCT06577857
Title: Minimally Invasive Micro Sclerostomy (MIMS®) Inferonasal Procedure: Long-Term Follow-Up Extension Study
Brief Title: Inferonasal MIMS® Procedure: Long-Term Follow-Up Extension Study
Status: Recruiting | Type: Observational
Sponsor: Sanoculis Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: MMS-EEU-8
Record Dates: First submitted 2024-08-27; First posted 2024-08-29 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Open Angle Glaucoma
Keywords: Intraocular Pressure; MIMS; Inferonasal; Minimally Invasive Glaucoma Surgery; Trabeculectomy; Sclerostomy; MIGS
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Inferonasal MIMS Surgery Cohort: Cohort that includes subjects that have undergone the MIMS® inferonasal surgery.
  Interventions: Device: Inferonasal Minimally Invasive Micro Sclerostomy

INTERVENTIONS:
Device: Inferonasal Minimally Invasive Micro Sclerostomy — The Inferonasal MIMS® procedure uses the proprietary MIMS® device, which creates a sclerostomy in the inferonasal quadrant of the eye.
  Other Names: Inferonasal MIMS

SUMMARY:
A long-term (24 and 30 months) follow-up extension, prospective, non-interventional, open label study for data collection from subjects who underwent prior MIMS® inferonasal surgery, in continuation of the previous clinical investigation with the MIMS® Device (MMS-EEU-5).

ELIGIBILITY:
Inclusion Criteria:

1. Subject who underwent MIMS® inferonasal procedure, and surgery was performed not earlier than 24 months from enrollment

Ages: 40 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population consists of subjects of Armenian descent that underwent the MIMS® inferonasal procedure, and surgery was performed not earlier than 24 months from enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 53 (Estimated)
Dates: Start 2022-11-04 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Intraocular Pressure Change (Baseline to 24 months) | Baseline to 24 months post-MIMS® surgery
  Change in IOP from medicated baseline to 24 months post-MIMS® surgery
Intraocular Pressure Change (Baseline to 30 months) | Baseline to 30 months post-MIMS® surgery
  Change in IOP from medicated baseline to 30 months post-MIMS® surgery
Change in Number of Topical Intraocular Pressure Lowering Medications (Baseline to 24 Months) | Medicated baseline to 24 months post-MIMS® surgery
  Change in the number of topical IOP-lowering medications from medicated baseline to 24 months post-MIMS® surgery
Change in Number of Topical Intraocular Pressure Lowering Medications (Baseline to 30 Months) | Medicated baseline to 30 months post-MIMS® surgery
  Change in the number of topical IOP-lowering medications from medicated baseline to 30 months post-MIMS® surgery
Surgery Success Rate (24 months) | 24 months post-MIMS® surgery
  Success rate 24 months post-MIMS® surgery
Surgery Success Rate (30 months) | 30 months post-MIMS® surgery
  Success rate 30 months post-MIMS® surgery

SECONDARY OUTCOMES:
Postoperative Complication Safety Outcomes | Baseline to 30 months post-MIMS® surgery
  Late (greater than 12 months) postoperative complications
Interventional Safety Outcomes | Baseline to 30 months post-MIMS® surgery
  Late (greater than 12 months) postoperative interventions

CONTACTS AND LOCATIONS:
Locations (1):
- S. Malayan Eye Center, Yerevan, Armenia

IPD SHARING:
Plan to Share IPD: Undecided